CLINICAL TRIAL: NCT00561873
Title: Phase-II-Study of Efficacy of OSAG 101 (Theraloc®) for Adolscent Patients With Recurrent High Grade Glioma
Brief Title: Nimotuzumab in Children With HGG
Status: Completed | Type: Observational
Sponsor: Oncoscience AG (Industry)
Collaborators: Children's Medical Hospital, University of Bonn, Germany (Other); University of Wuerzburg (Other); University of Bonn (Other); Dept. of Statistics, University of Dortmund, Germany (Other); CRM Biometrics GmbH (Industry); Heinrich-Heine University, Duesseldorf (Other); University Hospital Augsburg (Other); Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other); Children's Medical Hospital, University of Homburg/Saar, Homburg/Saar, Germany (Other); Children's Medical Hospital, Medical School Hannover, Hannover, Germany (Unknown); Children's Medical Hospital, University of Essen, Essen, Germany (Other); Dept. of Neuropediatrics and Muscle Disorders, University of Freiburg, Germany (Other); University of Cologne (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Regensburg (Other)
Other Study IDs: BN001-PED04
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: High Grade Glioma
Keywords: astrocytoma, glioblastoma, intrinsic pontine glioma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Determination of efficiency of nimotuzumab in children with high grade glioma.

DETAILED DESCRIPTION:
High grade malignant gliomas are tumors grade III and IV according to WHO classification, that originate from oligodendroglia and astrocytes, where the latter are also known as anaplastic astrocytoma(WHO grade III) and glioblastoma(WHO grade IV). This also includes intrinsic pontine gliomas of adolescents, which are usually not documented histologically due to their localisation, but they have a similar clinical progress when compared to high grade malignant astrocytic tumors. Among various molecular alterations, malignant gliomas overexpress EGFR (epidermal growth factor) in nearly 50% of cases, which is particularly pronounced in glioblastoma.(Schlegel 2003) Standard therapy consists of radical surgery as extensive as medically responsible followed by radiotherapy dose of 60 Gy, which is aimed at the area with a safety margin. The long-term efficacy of additional chemotherapy has been a subject for controversy for several decades. The combination of all three treatment modalities in grade III tumors can lead to median survival times of 3-5 years in adults.

For this treatment group reports of 5 year recurrence free periods in 33-50% of cases have been reported in children and adolescents.

For glioblastoma(WHO grade IV) 5year recurrence free periods are 3% in elderly patients and 10-20% for adolescents.(Schlegel 2003) In German speaking territories chemotherapy with Cisplatin, Etoposid and Ifosfamid is used as a postoperative treatment option for adolescents and this disease.(Wolff HIT-GBM) In case of recurrence therapy choices are even more limited, thus if medically feasible the enrolment in clinical trials is an option.

In this study the aim is to use an antibody directed against the EGF-receptor to effect the proliferation of the tumor cells negatively. Pilot studies conducted in adults indicate that the median survival time for patients with malignant glioma can be prolonged by the antibody treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of high grade glioma (WHO III und IV) [not needed for intrinsic pontine glioma]
* Progressive patients under primary therapy or first and second radiologically confirmed recurrence(MRI not older than 2 weeks) of high grade gliomas between the age of > 3 years < 20 years
* Lack of curative standard therapy which is currently under investigation in a national GPOH-therapy optimization study
* Sufficient haematological, renal and hepatic function (CTC Grad ≤ 2)
* Disease measurable radiologicaly in at least one dimension
* Life expectancy > 4 Weeks
* Written declaration of consent of the parents/legal guardians and if possible of the child after prior information

Exclusion Criteria:

* Curative therapy with an alternative method after diagnosis of progression and during this study
* Prior administration of human or murine antibody
* Pregnancy in girls of child-bearing age

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children, adolescents
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2004-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response rate according to RECIST criteria | week 8, week 21

SECONDARY OUTCOMES:
Progress free interval, Toxicity according to CTC criteria, Symptom control | week 8, week 21

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bode, Prof. MD, Principal Investigator — University Bonn
Locations (1):
- University Bonn, Children's Medical Hospital, Bonn, Germany

REFERENCES:
- See also: Related Info — http://ukb.uni-bonn.de